CLINICAL TRIAL: NCT04591938
Title: Safety and Efficacy of the FANTOM ENCORE Sirolimus-eluting Bioresorbable Scaffold for Treatment of De-novo Coronary Artery Disease: the ENCORE-I Study
Brief Title: FANTOM ENCORE Sirolimus-eluting Bioresorbable Scaffold for Treatment of De-novo CAD: the ENCORE-I Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Joost Daemen (Other)
Collaborators: Horizon 2020 - European Commission (Other); REVA Medical, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Joost Daemen, Interventional Cardiologist, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ENCORE-I
Record Dates: First submitted 2020-10-06; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Percutaneous Coronary Intervention; Myocardial Revascularization; Tomography, Optical Coherence
Keywords: Bioresorbable scaffold; Percutaneous Coronary Intervention; OCT

STUDY DESIGN:
Intervention Model Description: Prospective, multicentre, non-randomized, investigator-initiated study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other): Fantom Encore Bioresorbable scaffold implantation
  Interventions: Device: Fantom Encore Bioresorbable scaffold implantation

INTERVENTIONS:
Device: Fantom Encore Bioresorbable scaffold implantation — Fantom Encore Bioresorbable scaffold implantation

SUMMARY:
Prospective, multicentre, non-randomized, investigator-initiated study aiming to assess the safety and efficacy of the Fantom Encore sirolimus-eluting bioresorbable scaffold (BRS).

DETAILED DESCRIPTION:
Up to 50 consecutive participants with de-novo non-complex obstructive coronary lesions and non-ST elevation acute coronay syndromes or stable angina pectoris will be included in the Netherlands and Belgium.

Device performance and behaviour will be assessed by angiography and optical coherence tomography at the index procedure and at 13 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Stable angina, unstable angina or documented silent ischemia (invasive or non-invasive test) or non-ST segment elevation acute myocardial infarction.
* De-novo non-complex coronary obstructive lesions (>50% stenosis as assessed by quantitative coronary analysis (QCA))
* The patient is willing and able to comply with the specified follow-up evaluations.
* Reference vessel diameter (RVD) ≥ 2.5 mm and ≤ 4.0 mm by QCA.
* During pre-dilatation, the pre-dilatation balloon is uniformly expanded to the full intended diameter.
* Target segment suitable for OCT imaging

Exclusion Criteria:

* Target vessel with a distal Thrombolysis In Myocardial Infarction (TIMI) flow 0 or 1.
* Target lesion located within 5.0 mm of vessel origin.
* Lesion type ACC/AHA C.
* Heavily calcified lesion
* Severe tortuosity
* Target lesion is located in or supplied by an arterial or venous bypass graft.
* Target lesion requires treatment with a device other than the pre-dilatation balloon prior to scaffold placement (including but not limited to directional coronary atherectomy, excimer laser, rotational atherectomy, etc.).
* Unsuccessful pre-dilatation, defined as a residual diameter stenosis ≥ 30%, assessed by QCA.
* Planned future revascularization of non-culprit lesions.
* Presence of another device (stent or scaffold) located within the same segment (5mm from the target lesion borders).
* Patient is currently participating in another study with an investigational device or an investigational drug and has not completed the entire follow-up period.
* Impaired renal function (eGFR <30ml/min).
* Patient has a contraindication for the use of double antiplatelet therapy for at least 12 months.
* Pregnant or breastfeeding patients.
* Patient has a known allergy to contrast medium, sirolimus, Tyrosine-derived polycarbonate or other structurally related compounds.
* Patient is receiving chronic oral or intravenous immunosuppressive therapy or has known life-limiting immunosuppressive or autoimmune disease (diabetes mellitus is not an exclusion criteria).
* Patient has a co-morbidity, which reduces life expectancy to ≤ 24 months, or social-economic factors making compliance with the study requirements difficult.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Device-Oriented Composite Endpoint (DOCE) | 12 months
  A composite of cardiac death, target vessel-related non-fatal myocardial infarction (MI) and clinically-driven target lesion revascularization(CD-TLR).

SECONDARY OUTCOMES:
Subcomponents of DOCE | 30 days, 6, 12, 24, 36, 48 and 60 months
  Subcomponents of the Device-Oriented Composite Endpoints
Target vessel revascularization (TVR) | 30 days, 6, 12, 24, 36, 48 and 60 months
  Target vessel revascularization
Definite or probable stent thrombosis (ST) | 30 days, 6, 12, 24, 36, 48 and 60 months
  Stent thrombosis

OTHER OUTCOMES:
Angiographic outcomes at baseline | 0 days
  Acute gain
Angiographic outcomes at baseline | 0 days
  acute recoil
Angiographic outcomes at baseline | 0 days
  Incidence of procedural complications (dissection >B, perforation, vessel closure, slow flow or no-reflow, intra-procedure scaffold thrombosis)
Angiographic outcomes at follow-up | 13 months
  In-device and in-segment late lumen loss (LLL)
Angiographic outcomes at follow-up | 13 months
  In-device and in-segment binary restenosis rate
Device performance | 0 days
  Device success
Device performance | 0 days
  Procedural success
Optical coherence tomography outcomes at baseline | 0 days
  Incomplete strut apposition (ISA)
Optical coherence tomography outcomes at baseline | 0 days
  Scaffold expansion
Optical coherence tomography outcomes at baseline | 0 days
  Scaffold eccentricity
Optical coherence tomography outcomes at baseline | 0 days
  Scaffold symmetry index
Optical coherence tomography outcomes at baseline | 0 days
  Edge dissection
Optical coherence tomography outcomes at baseline | 0 days
  In-device and in-segment endothelial shear stress
Optical coherence tomography outcomes at follow-up | 13 months
  Neointima thickness
Optical coherence tomography outcomes at follow-up | 13 months
  Percentage of patent struts
Optical coherence tomography outcomes at follow-up | 13 months
  Percentage of uncovered struts
Optical coherence tomography outcomes at follow-up | 13 months
  Persistent ISA
Optical coherence tomography outcomes at follow-up | 13 months
  Acquired ISA
Optical coherence tomography outcomes at follow-up | 13 months
  Scaffold eccentricity index
Optical coherence tomography outcomes at follow-up | 13 months
  Scaffold symmetry index
Optical coherence tomography outcomes at follow-up | 13 months
  In-device and in-segment late lumen area loss
Optical coherence tomography outcomes at follow-up | 13 months
  In-device and in-segment binary restenosis rate.
Optical coherence tomography outcomes at follow-up | 13 months
  In-device and in-segment endothelial shear stress

CONTACTS AND LOCATIONS:
Overall Officials: Joost Daemen, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (3):
- Belgium (2):
  - Ziekenhuis Oost-Limburg, Genk
  - Universitair Ziekenhuis Leuven, Leuven
- Erasmus Medical Center, Rotterdam, Netherlands